CLINICAL TRIAL: NCT04897763
Title: A Pilot Open-label, Feasibility Study to Assess safEty, Tolerability, Radiation Dosimetry, and Imaging Properties of 89Zr-labeled giRenTuximab (89Zr-Girentuximab) in patIents With Non-musclE-iNvasive Bladder CancEr (NMIBC)
Brief Title: Assessment of Safety, Tolerability, Radiation Dosimetry, Imaging Properties of 89Zr-girentuximab in Patients With NMIBC
Acronym: PERTINENCE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: ATONCO (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICO-2021-03
Record Dates: First submitted 2021-05-17; First posted 2021-05-24 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer
Keywords: Non-muscle-invasive bladder cancer (NMIBC); 89Zr-Girentuximab PET; pilot study; 89Zr-TLX250 PET; carbonic anhydrase IX (CAIX)
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Monocentric, open prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-TLX250 (Experimental): 89Zr-TLX250 (89Zr-girentuximab) PET/CT performed for all aptients
  Interventions: Drug: 89Zr-TLX250

INTERVENTIONS:
Drug: 89Zr-TLX250 — 89Zr-TLX250 (89Zr-girentuximab) PET/CT performed for all aptients
  Other Names: [89Zr]Zr-girentuximab

SUMMARY:
The purpose of this study is to evaluate the use of 89Zr-labeled girentuximab (89Zr-TLX250) as a novel, carbonic anhydrase IX (CAIX) targeted PET/CT radiopharmaceutical for the imaging of Non-muscle-invasive bladder cancer (NMIBC) patients.

DETAILED DESCRIPTION:
There is a real need for treatment of NMIBC. Currently, treatment options include Bacillus Calmette-Guerin (BCG) intravesical immunotherapy and mitomycin C chemotherapy. These therapies are efficient for some time but relapses repeat them at more and more close intervals and finally patients are refractory to them and require a radical cystectomy.

CAIX is expressed in 70% to 90% of bladder cancers but not in normal urothelial tissue. CAIX is expressed on the membrane of Non-Muscle-Invasive Bladder Cancer cells.

Girentuximab, an anti-CAIX antibody could be a promising target in NMIBC. PET/CT with Girentuximab labelled with 89Zirconium will be used for diagnosis purpose. 89Zr-Girentuximab will be administered by intravesical instillation.

In this study, patients with Non-Muscle-Invasive Bladder Cancer (NMIBC) will be enrolled in this study after confirmation of their eligibility.

A single intravesical administration of 89Zr-Girentuximab will be performed at day 0.

Multiple PET/CT imaging sessions will be performed on day 0, day 1 and day 2 in order to evaluate the bladder and the whole body 89Zr girentuximab uptake.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Female or male, Age ≥ 18 years at time of study entry.
* Performance Status: 0 or 1.
* Clinical evidence of NMIBC based on cystoscopy and proven histologically of papillary tumors.
* Histologically-confirmed pTa Grade 3 or pT1 Grade 3 bladder cancer patients relapsing without muscle invasion.
* Negative sterile Urine cytobacteriological testing at baseline (T0).
* Consent to use a contraception method for at least 30 days after administration of 89Zr-girentuximab.
* Patient has valid health insurance.

Exclusion Criteria:

* Patient with urinary incontinence.
* Known hypersensitivity to girentuximab.
* Exposure to any experimental diagnostic or therapeutic drug within 30 days prior the date of planned administration of 89Zr-girentuximab
* Exposure to any radiopharmaceutical within 30 days (corresponding to 10 half-lives of Zr-89) prior to the administration of 89Zr-girentuximab
* Patients suffering from a bladder cancer at stage pT2, pT3 or pT4
* Serious non-malignant disease that may interfere with the objectives of the study or with the safety or compliance of the patient; as judged by the investigator
* Concomitant cancer in the past 5 years except cutaneous cancers (except melanoma) and in situ carcinoma
* Prior chemotherapy, radiotherapy (other than short cycle of palliative radiotherapy), immunotherapy within 21 days of 89Zr-girentuximab administration
* Patients with known human immunodeficiency viruses (HIV), Hepatitis B virus (HBV) and Hepatitis C Virus (HCV) infections,
* Pregnant or likely to be pregnant or nursing patient.
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study
* Persons deprived of their liberty, under a measure of safeguard of justice, under guardianship or placed under the authority of a guardian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline ROUSSEAU, MD, PhD, Study Chair — Institut de Cancerologie de l'Ousest - ICO
Locations (1):
- Institut de cancerologie de l'Ouest, Saint-Herblain, France

REFERENCES:
- See also: PubMed — https://pubmed.ncbi.nlm.nih.gov/40227816/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start date First patient was enrolled: 15 DEC 2021 End of trial date (last visit of last patient): 26 SEP 2022
Pre-assignment Details: All screened patients have been enrolled
Groups:
- 89Zr-TLX250 PET/CT: 89Zr-TLX250 (89Zr-girentuximab) PET/CT performed for all patients after 89Zr-TLX250 (89Zr-girentuximab) administration
Period: Overall Study
Arm/Group | 89Zr-TLX250 PET/CT
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 89Zr-TLX250: 89Zr-TLX250 (89Zr-girentuximab) PET/CT performed for all patients after 89Zr-TLX250 (89Zr-girentuximab) administration
Arm/Group | 89Zr-TLX250
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  France | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Uptake Spot in 89Zr-girentuximab PET/CT Images
Description: The presence or absence of uptake spot in bladder wall of 89Zr-girentuximab bladder and whole body PET/CT Images.
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Groups:
- 89Zr-TLX250 (89Zr-girentuximab) PET/CT: 89Zr-TLX250 (89Zr-girentuximab) PET/CT performed for all patients after 89Zr-TLX250 (89Zr-girentuximab) administration
Arm/Group | 89Zr-TLX250 (89Zr-girentuximab) PET/CT
Number analyzed (Participants) | 6
Participants
  Uptake spot in bladder wall with early recurrence | 1
  Uptake spot in bladder wall with post-TURB inflammatory scarring reaction | 2
  No uptake spot in bladder wall | 3

2. Primary Outcome: Number of Patients With Positive and Negative 89Zr-girentuximab Blood Dosing
Description: 89Zr-girentuximab activity dosing in blood is measured. The number of patients with Positive and negative 89Zr-girentuximab Blood dosing is evaluated.
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | 89Zr-TLX250 (89Zr-girentuximab) PET/CT
Number analyzed (Participants) | 6
Participants
  Positive 89Zr-girentuximab Blood dosing | 1
  Negative 89Zr-girentuximab Blood dosing | 5

3. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Serious adverse events, related or not to 89Zr-girentuximab, are assessed up to Day 30 after 89Zr-girentuximab administration, using CTC-AE scale version 5.0
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 89Zr-TLX250 (89Zr-girentuximab) PET/CT
Number analyzed (Participants) | 6
Participants
  Urinary retention grade 2 not related to 89Zr-TLX250 (89Zr-girentuximab) PET/CT | 1
  Haemorrhage grade 3 not related to 89Zr-TLX250 (89Zr-girentuximab) PET/CT | 1
  No SAE | 4

4. Secondary Outcome: Number of Patients With Positive and Negative CA-IX Expression in Tumor Cells
Description: The expression of CAIX is by immunohistochemistry in tumor sample from TransUrethral Resection of Bladder Tumor (TURBT) or cystectomy
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | 89Zr-TLX250 (89Zr-girentuximab) PET/CT
Number analyzed (Participants) | 6
Participants
  Positive CA-IX expression in tumor cells | 5
  Negative CA-IX expression in tumor cells | 1

5. Secondary Outcome: Number of Participants With Adverse Events Related to 89Zr-girentuximab
Description: Adverse events related to 89Zr-girentuximab are assessed up to Day 3 After 89Zr-girentuximab Administration, using CTC-AE scale version 5.0
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | 89Zr-TLX250 (89Zr-girentuximab) PET/CT
Number analyzed (Participants) | 6
Participants
  Urethral bleeding grade 1 not related to 89Zr-TLX250 (89Zr-girentuximab) PET/CT | 1
  No adverse events | 5

6. Secondary Outcome: Radiation Protection Management
Description: Radiation exposure of 3 staff membres (extremities and Whole body: µSv). A value greater than 4mSv is considered abnormal.
Time Frame: 3 days
Population: Assessments were conducted on three staff members involved in the administration of 89Zr-TLX250 (89Zr-girentuximab) to determine the presence or absence of staff contamination from the administered radioactivity during patient management.
Measure: Mean (Full Range); unit: µSv
Arm/Group | 89Zr-TLX250 (89Zr-girentuximab) PET/CT
Number analyzed (Participants) | 3
µSv
  Whole body radiation exposure of staff | 5.5 [1 to 10]
  Extremities radiation exposure of staff | 5 [0 to 10]

7. Secondary Outcome: Radiation Protection Management
Description: Radiopharmaceutical management from intravesical instillation to elimination (surfasic contamination measured in counts/second).
Time Frame: 1 day
Population: Measurement of radioactivity on the urinary catheter, cotton swabs, diapers, and gloves to assess potential radioactivity contamination.
Measure: Mean (Full Range); unit: counts per second
Units Other Than Participants: Materials exposed to radioactivity
Arm/Group | 89Zr-TLX250 (89Zr-girentuximab) PET/CT
Number analyzed (Participants) | 6
Number analyzed (Materials exposed to radioactivity) | 4
counts per second | 115 [50 to 180]

ADVERSE EVENTS:
Time Frame: From the date of administration of 89Zr- Girentuximab until 30 days after administration
Arm/Group | 89Zr-TLX250
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 89Zr-TLX250 (N=6)
Urinary retention (Renal and urinary disorders) | 1 (1) — Urinary retention grade 2, not related to investigational product, hospitalisation from 22 FEB 2022 to 23 FEB 2022
Bladder bleeding (Renal and urinary disorders) | 1 (1) — Bladder bleeding following a Transurethral Resection of Bladder Tumor, grade 3, not related to investigational product
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 89Zr-TLX250 (N=6)
Urethral bleeding (Renal and urinary disorders) | 1 (1) — Urethral bleeding grade 1, not related to investigational product

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT04897763/Prot_SAP_000.pdf